CLINICAL TRIAL: NCT04662944
Title: A Non-interventional Study to Assess the Influence of Automated Optical Coherence Tomography (OCT) Image Enrichment With Segmentation Information on Disease Activity Assessment in Patients Treated With Licensed Anti- VEGF Injections
Brief Title: A Non-interventional Study to Assess the Influence of Automated Optical Coherence Tomography Image Enrichment With Segmentation Information on Disease Activity Assessment in Patients Treated With Licensed Anti- VEGF Injections
Acronym: RAZORBILL
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A2402
Record Dates: First submitted 2020-11-24; First posted 2020-12-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: nAMD; Neovascular Age-Related Macular Degeneration; anti-VEGF; RAZORBILL; optical coherence tomography; OCT; Artificial Intelligence; Machine learning; Automatic OCT segmentation
MeSH Terms: interventions — brolucizumab; Ranibizumab; aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Licensed anti-VEGFs: Patients being treated for nAMD with licensed anti-VEGFs
  Interventions: Drug: brolucizumab; Drug: ranibizumab; Drug: aflibercept

INTERVENTIONS:
Drug: brolucizumab — There was no treatment allocation. Patients administered Brolucizumab by prescription that started before inclusion of the patient into the study were enrolled.
Drug: ranibizumab — There was no treatment allocation. Patients administered Ranibizumab by prescription that started before inclusion of the patient into the study were enrolled.
Drug: aflibercept — There was no treatment allocation. Patients administered Aflibercept by prescription that started before inclusion of the patient into the study were enrolled.

SUMMARY:
RAZORBILL was an observational, multicenter, multinational, open-label, study designed primarily to investigate the influence of automated OCT image enrichment with segmentation information on disease activity assessment in nAMD patients treated with licensed anti-VEGFs

DETAILED DESCRIPTION:
The main goal of this study was to assess to what degree disease activity assessment is influenced and supported by the enrichment of OCT images with segmentation information (i.e. by identification, highlighting and quantification of pathological fluid compartments associated with neovascular activity).

The study comprised a prospective data collection phase and a retrospective analysis of OCT images phase. The prospective observation period per patient was up to 12 months.

The study included patients (naïve patients and patients who had been pre-treated with licensed anti-VEGFs not more than 3 years) being treated for nAMD with brolucizumab, ranibizumab, or aflibercept according to the respective drug label.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nAMD
* Male and Female patients with ≥18 years of age at index
* Receipt of at least one injection of brolucizumab, ranibizumab or aflibercept during the recruitment period
* Signed written informed consent
* Patients for whom a therapy with brolucizumab, ranibizumab or aflibercept is medically indicated according to the respective label
* Intraretinal and/or subretinal fluid affecting the central subfield of the study eye at screening

Exclusion Criteria:

* Patients treated for any other retinal disease than nAMD within 6 months prior to the index date (e.g. patients treated for retinal vein occlusion, diabetic macular oedema, myopic CNV, and have diagnoses of diabetes-related macular degeneration)
* Central subfield of the study eye affected by fibrosis or geographic atrophy or total area of fibrosis >50% of the total lesion in the study eye at screening
* Any active intraocular or periocular infection or active intraocular inflammation in either eye at index date
* Patients who have been on anti-VEGF treatment for longer than 3 years (before index date)
* Patients who have any contraindication and are not eligible for treatment with the chosen anti-VEGF treatment as according to the respective label.
* Any medical or psychological condition, in the treating physician's opinion, which may hinder the patient from participating in this study for the expected 12 months
* Patients participating, in parallel, in an interventional clinical trial
* Patients participating, in parallel, in any other Novartis sponsored NIS generating primary data for an anti-VEGF drug

Ages: 18 Years to 199 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects being treated for nAMD with brolucizumab, ranibizumab, or aflibercept according to the respective drug label.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Odds ratio of disease activity assessment from Optical Coherence Tomography (OCTs) with and without enrichment | 12 months
  An odds ratio of disease activity assessment from OCTs with and without enrichment was reported with a 95% confidence interval.
Degree of agreement in classification of disease activity using enriched and non-enriched OCT images | 12 months
  Degree of agreement in classification of disease activity assessed by Krippendorff's alpha using OCT images

SECONDARY OUTCOMES:
Difference in time needed for Disease Activity Assessment (DAA) between reviews with and without enrichment | 12 months
  the difference in time to DAA (time between begin of OCT viewing and result sub-mission) between cases reviewed with and without use of segmentation information was calculated.
Difference in confidence in DAA between reviews with and without enrichment | 12 months
  difference in confidence in DAA between cases reviewed with and without enrichment (rating of 1-10 per case, whereby a rating of 10 meant maximal confidence) was calculated
Acceptance of Discovery by physicians and whether it can optimize the ophthalmic clinical workflow | Month 12
  Physicians used a digital solution Discovery for managing imaging data and automatic segmentation of OCT volumes. To understand if such a tool is well suited for its role in its current form, holds value for physicians and can optimize clinical workflow, physicians were invited to complete questionnaires regarding their user experience.
Percentage of patients with absence of Subretinal Fluid, Intraretinal Fluid and Pigment Epithelium Detachment | Month 12
  Percentage of patients with absence of Subretinal Fluid, Intraretinal Fluid and Pigment Epithelium Detachment was provided
Central Subfield Thickness (CST) change | 12 months
  Course of Central Subfield Thickness (CST) change was provided
Best-corrected visual acuity change from baseline | 12 months
  Best-corrected visual acuity change from baseline was provided
Percentage of patients with ocular and non-ocular adverse events | 12 months
  Percentage of patients with ocular and non-ocular adverse events was provided
Subjective assessment of system correctness | 12 months
  Investigators assessed the correctness of the system on a scale from 0 to 10 (10 corresponds to maximum correctness) if segmentation algorithm was used.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Canada (3):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Germany (6):
  - Novartis Investigative Site, Ludwigsburg, Baden-Wurttemberg
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Ireland (2):
  - Novartis Investigative Site, Glasnevin, Dublin 9
  - Novartis Investigative Site, Waterford
- Novartis Investigative Site, Milan, MI, Italy
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Bormujos, Sevilla
  - Novartis Investigative Site, León

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258A2402 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18187